CLINICAL TRIAL: NCT03883048
Title: The Optimal Noninvasive Indicator for Identify Pulmonary Hypertension Will be Determined. Difference of Some Indexes Between Bronchiectasis With Pulmonary Hypertension and Bronchiectasis Without Pulmonary Hypertension.
Brief Title: Idiopathic Bronchiectasis and Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Proffessor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2018052395
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Bronchiectasis; Pulmonary Hypertension
MeSH Terms: conditions — Bronchiectasis; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation of bronchiectasis with pulmonary hypertension

SUMMARY:
Patients with idiopathic bronchiectasis who received right heart catheterization (RHC) were included to evaluate the consistency between pulmonary arterial pressure (PAP) and other noninvasive indicators (pulmonary arterial systolic pressure [PASP] calculated by echocardiography, main pulmonary artery [MPA] diameter and MPA/ascending aorta ratio on chest high-resolution computed tomography [HRCT]). Then the optimal noninvasive indicator for identify PH was determined and its critical point was obtained according to the Youden Index. Based on this, we investigate the proportion, risk factors and prognosis of PH in idiopathic bronchiectasis patients in another large-scale population.

DETAILED DESCRIPTION:
Between April 2011 and December 2019, the data of idiopathic bronchiectasis patients were analyzed to determine the optimal noninvasive tool to identify PH. Based on the patients who received RHC examination, Spearman correlation was used to assess the correlation between mean pulmonary arterial pressure (mPAP) and systolic pulmonary arterial pressure (sPAP) measured by RHC and other noninvasive indicators (estimated PASP assessed by echocardiography, main pulmonary artery (MPA) diameter and MPA/ ascending aorta (AA) ratio on chest HRCT scan), in order to screening out the optimal indicator to identify PH. Then the sensitivity and specificity of the indicator was calculated through the receiving operating characteristics (ROC) analysis and the critical point of the indicator was determined by Youden index.

Based on critical point of that indicator, a large sample study from hospital medical database for patients with idiopathic bronchiectasis in Shanghai Pulmonary Hospital (Shanghai, China) between May 2013 and December 2019 was conducted. The following data were collected: demographic information (i.e., age and sex); clinical characteristics (age of symptom onset, duration after bronchiectasis diagnosis, and body mass index [BMI]); radiological presentation (the type of bronchiectasis, and involved lung lobe and segment); pulmonary function (forced vital capacity [FVC], forced expiratory volume in 1 second [FEV1], and FEV1/FVC); N-terminal pro brain natriuretic peptide (N-proBNP); arterial blood gas and microbiological detection in respiratory tract specimen (sputum or bronchoalveolar lavage fluid). The number of hospitalizations and emergency visits in past 12 months before the first hospitalization were collected based on patient's medical records. Patients were followed up by telephone until December 2021.

The idiopathic patients who received echocardiography examination were divided into two groups. The risk factors of PH associated with idiopathic bronchiectasis and the effect of PH on the prognosis of patients with bronchiectasis were analyzed through statistical method.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18;
2. Patients with typical bronchiectasis on CHEST HRCT;
3. Patients with bronchiectasis without known cause.

Exclusion Criteria:

1. Patients with allergic bronchopulmonary aspergillosis (ABPA).
2. Patients with bronchiectasis combined with pulmonary tuberculosis and non-tuberculous mycobacterium tuberculosis.
3. Patients with bronchiectasis due to genetic factors.
4. Bronchiectasis patients with connective tissue diseases.
5. Patients with bronchiectasis with interstitial lung disease.
6. Combined with pulmonary embolism, pneumothorax, mediastinal emphysema and lung tumor.
7. Patients with bronchiectasis associated with chronic obstructive pulmonary and bronchial asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Between April 2011 and December 2019, patients with bronchiectasis received right heart catheterization examination.
  2. The patients with idiopathic bronchiectasis received echocardiography from May 2013 to Dec 2019.
Sampling Method: Non-Probability Sample
Enrollment: 1606 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The optimal noninvasive indicator for identify pulmonary hypertension | April/01/2011-Decemeber/31/2019
  Based on the patients who received right heart catheterization examination, the optimal noninvasive indicator for identify PH was determined
Differance of some indexes between Bronchiectasis with pulmonary hypertension and Bronchiectasis without pulmonary hypertension | May/01/2013-Decemeber/31/2019
  Differance of some indexes (ie. course, clinical presentation, type and scope of bronchiolitis, lung function, pseudomonas aeruginosa in respiratory tract specimen and prognosis) between Bronchiectasis with pulmonary hypertension and Bronchiectasis without pulmonary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Mr Xu, Doctor, Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided